CLINICAL TRIAL: NCT03343340
Title: Early Versus Late CRRT (Continuous Renal Replacement Therpay) in ACLF (Acute on Chronic Liver Failure) Patients With Septic Shock and AKI (Acute Kidney Injury) - A Randomized Controlled Trial
Brief Title: Early Versus Late CRRT in ACLF Patients With Septic Shock and AKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-CRRT-01
Record Dates: First submitted 2017-09-23; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-09

CONDITIONS: Septic Shock and Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early CRRT (Experimental): Early Continous Renal Replacement Therapy within 6 hours + Standard Medical Therapy
  Interventions: Other: Early CRRT; Other: Standard Medical Therapy
- Late CRRT (Active Comparator): Late Continous Renal Replacement Therapy + Standard Medical Therapy
  Interventions: Other: Late CRRT; Other: Standard Medical Therapy

INTERVENTIONS:
Other: Early CRRT — Continous Renal Replacement Therapy
  Arms: Early CRRT
Other: Late CRRT — Continous Renal Replacement Therapy
  Arms: Late CRRT
Other: Standard Medical Therapy — Standard Medical Therapy

SUMMARY:
Consecutive patients with ACLF (Acute on Chronic Liver Failure) and septic shock with AKI (Acute Kidney Injury) who give written informed consent will be included in this prospective trial at ILBS. At baseline s, endotoxin levels, NT-Pro BNP, , urine N-GAL will be done for all patients. A 10 ml serum sample will be stored for doing a cytokine profile. Septic shock will be defined by the presence of two or more diagnostic criteria for the systemic inflammatory response syndrome, proven or suspected infection with hypotension non-responsive to adequate fluid resuscitation assessed by no evidence of stroke volume variation on flow track and need of a vasopressor to achieve a target mean arterial pressure (MAP) of ≥ 65 mm Hg. A record of CVP, IVC diameter and B-lines on ultrasound lung would also be done. Patients with age less than 18 years, severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD) pregnancy, chronic kidney disease, patients already meeting emergency criteria for immediate hemodialysis at the time of randomization as specified in the late group, patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit, extremely moribund patients with an expected life expectancy of less than 24 hours, failure to give informed consent from family members.

ELIGIBILITY:
Inclusion Criteria:

- Patients with ACLF defined based on APASL criteria with septic shock associated AKI

Exclusion Criteria:

* Patients with age less than 18 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
* Pregnancy
* Chronic kidney disease on hemodialysis
* Patients with Hepatorenal Syndrome, post renal obstructive AKI, AKI due to glomerulonephritis, interstitial nephritis or vasculitis
* Patients already meeting emergency criteria for immediate hemodialysis at the time of randomization as specified in the late group (serum potassium>6 meq/lt, metabolic acidosis ph<7.12, acute pulmonary edema, severe volume overload with hypoxemia non-responsive to diuretic treatment)
* Patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Hemodynamic instability requiring very high dose of vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-09-25 (Estimated); Study Completion 2018-09-25 (Estimated)

PRIMARY OUTCOMES:
Transplant Free Survival | 28 days

SECONDARY OUTCOMES:
Incidence of intradialytic hypotension i.e. defined as a decrease in systolic blood pressure by ≥20 mm Hg or a decrease in MAP by 10 mm Hg associated with symptoms | 1 year
Hemodynamic stability i.e. maintenance of MAP on dialysis without increase in the vasopressors | 1 year
Dialysis efficiency as measured by Urea Reduction ratio at 48 hours | 2 days
Achievement of target ultrafiltration goals | 1 year
Recovery in renal functions defined as an increase in urine output to more than 400 ml/day | 1 year
Duration of mechanical ventilation and ICU (Intensive Care Unit) stay | 1 year
Improvement in SOFA (Sequential Organ Failure Assessment ) ( by 2 points) scores | 1 year
Improvement in APACHE (Acute Physiology and Chronic Health Evaluation) ( by 2 points) scores | 1 year
Improvement in MELD (Model for End Stage Liver Disease) ( by 2 points) scores | 1 year
Improvement in lactic acidosis and lactate clearance at 6 hours after initiation of CRRT | within 6 hours
Improvement in lactic acidosis and lactate clearance at 12 hours after initiation of CRRT | within 12 hours
Improvement in lactic acidosis and lactate clearance at 24 hours after initiation of CRRT | within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787